CLINICAL TRIAL: NCT02791412
Title: Ten-Year Outcomes of Stents Versus Coronary-Artery Bypass Grafting for Left Main Coronary Artery Disease in Korea : Multicenter, Long-term, Observational Trial
Brief Title: Ten-Year Outcomes of Stents Versus Coronary-Artery Bypass Grafting for Left Main Coronary Artery Disease
Acronym: MAIN COMPARE
Status: Completed | Type: Observational
Sponsor: Seung-Jung Park (Other)
Collaborators: CardioVascular Research Foundation, Korea (Other)
Responsible Party: Sponsor-Investigator, Seung-Jung Park, professor of medicine, Asan Medical Center
Organization: Asan Medical Center (Other)
Other Study IDs: AMCCV2016-08
Record Dates: First submitted 2016-05-30; First posted 2016-06-06 (Estimated); Last update posted 2018-06-26 (Actual); Status verified 2018-06

CONDITIONS: Coronary Arteries
Keywords: left main; unprotected; percutaneous coronary intervention; coronary-artery bypass graft
MeSH Terms: interventions — Percutaneous Coronary Intervention; Coronary Artery Bypass

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- unprotected left main: undergone percutaneous coronary intervention or coronary artery bypass graft
  Interventions: Procedure: percutaneous coronary intervention or coronary-artery bypass graft

INTERVENTIONS:
Procedure: percutaneous coronary intervention or coronary-artery bypass graft

SUMMARY:
The purpose of this study is to evaluate long-term outcome of treatment(percutaneous coronary intervention or coronary-artery bypass graft) in unprotected left main coronary artery stenosis in Korea.

ELIGIBILITY:
Inclusion Criteria:

* Unprotected left main disease

Exclusion Criteria :

* No exclusion criteria

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergone percutaneous coronary intervention or coronary-artery bypass graft for treatment of unprotected left main disease
Sampling Method: Non-Probability Sample
Enrollment: 2240 (Actual)
Dates: Start 2017-01-13 (Actual); Primary Completion 2018-05-30 (Actual); Study Completion 2018-05-30 (Actual)

PRIMARY OUTCOMES:
composite event | 10 years
  all-cause death, myocardiac infarction, revascularization

CONTACTS AND LOCATIONS:
Locations (12):
- South Korea (12):
  - Asan Medical Center, Seoul, Songpa-gu
  - Kyungpook National University Hospital, Daegu
  - Chungnam National University Hospital, Daejeon
  - Chonnam National University Hospital, Gwangju
  - Gachon University Gil Hospital, Incheon
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Seoul
  - The Catholic University of Korea Seoul St. Mary's Hospital, Seoul
  - The Catholic University of Korea, Yeouido St. Mary's Hospital, Seoul
  - Seoul National University Bundang hospital, Sungnam
  - Ajou University Hospital, Suwon

IPD SHARING:
Plan to Share IPD: No
This is not a publicly funded trial.

REFERENCES:
- [Derived] Kim TO, Kang DY, Ahn JM, Kim MJ, Lee PH, Kim H, Choi Y, Lee J, Lee JM, Jo HH, Park YS, Lim SM, Park SJ, Park DW. Impact of Target Lesion Revascularization on Long-Term Mortality After Percutaneous Coronary Intervention for Left Main Disease. JACC Cardiovasc Interv. 2024 Jan 8;17(1):32-42. doi: 10.1016/j.jcin.2023.10.068. PMID 38199751
- [Derived] Yoon YH, Ahn JM, Lee JB, Kang DY, Park H, Jeong YJ, Lee J, Kim JH, Yang Y, Hyun J, Lee PH, Park DW, Park SJ. Time-Dependent Impact of Sex on the Long-Term Outcomes After Left Main Revascularization. J Am Heart Assoc. 2022 Mar;11(5):e021720. doi: 10.1161/JAHA.121.021720. Epub 2022 Feb 22. PMID 35189706
- [Derived] Kang DY, Ahn JM, Yun SC, Park H, Cho SC, Kim TO, Park S, Lee PH, Lee SW, Park SW, Park DW, Park SJ. Long-Term Clinical Impact of Intravascular Ultrasound Guidance in Stenting for Left Main Coronary Artery Disease. Circ Cardiovasc Interv. 2021 Oct;14(10):e011011. doi: 10.1161/CIRCINTERVENTIONS.121.011011. Epub 2021 Oct 19. PMID 34665659
- [Derived] Lee K, Ahn JM, Yoon YH, Kang DY, Park SY, Ko E, Park H, Cho SC, Park S, Kim TO, Lee PH, Lee SW, Park SW, Park DW, Park SJ. Long-Term (10-Year) Outcomes of Stenting or Bypass Surgery for Left Main Coronary Artery Disease in Patients With and Without Diabetes Mellitus. J Am Heart Assoc. 2020 Apr 21;9(8):e015372. doi: 10.1161/JAHA.119.015372. Epub 2020 Apr 20. PMID 32310027
- [Derived] Kim TO, Ahn JM, Kang DY, Kim SO, Park S, Park H, Lee PH, Lee SW, Park SW, Park DW, Park SJ. Rates and Independent Correlates of 10-Year Major Adverse Events and Mortality in Patients Undergoing Left Main Coronary Arterial Revascularization. Am J Cardiol. 2020 Apr 15;125(8):1148-1153. doi: 10.1016/j.amjcard.2020.01.023. Epub 2020 Jan 29. PMID 32085865
- [Derived] Yoon YH, Ahn JM, Kang DY, Park H, Cho SC, Lee PH, Lee SW, Park SW, Park DW, Park SJ. Impact of SYNTAX Score on 10-Year Outcomes After Revascularization for Left Main Coronary Artery Disease. JACC Cardiovasc Interv. 2020 Feb 10;13(3):361-371. doi: 10.1016/j.jcin.2019.10.020. PMID 32029254
- [Derived] Park DW, Ahn JM, Yun SC, Yoon YH, Kang DY, Lee PH, Lee SW, Park SW, Seung KB, Gwon HC, Jeong MH, Jang Y, Kim HS, Seong IW, Park HS, Ahn T, Chae IH, Tahk SJ, Park SJ. 10-Year Outcomes of Stents Versus Coronary Artery Bypass Grafting for Left Main Coronary Artery Disease. J Am Coll Cardiol. 2018 Dec 11;72(23 Pt A):2813-2822. doi: 10.1016/j.jacc.2018.09.012. Epub 2018 Sep 24. PMID 30261236